CLINICAL TRIAL: NCT04403906
Title: Evaluation of the PCL Rapid Point of Care Antigen Test for Severe Acute Respiratory Syndrome Coronavirus 2
Brief Title: Somerset and South Essex Coronavirus Antigen Testing
Acronym: SOCRATES
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Not yet recruiting
Sponsor: Somerset NHS Foundation Trust (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Diagnostic
Other Study IDs: IRAS283137
Record Dates: First submitted 2020-05-21; First posted 2020-05-27 (Actual); Last update posted 2020-05-27 (Actual); Status verified 2020-05

CONDITIONS: COVID; SARS-CoV 2
Keywords: Anitgen testing; Coronavirus
MeSH Terms: conditions — Coronavirus Infections

STUDY DESIGN:
Intervention Model Description: Evaluation of diagnostic test - point of care
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- PCL Rapid Antigen Test arm (Experimental): Single arm trial design. Only patients undergoing standard clinical testing (SARS-CoV-2 PCR test) and consenting for additional testing with the PCL rapid antigen test will be included
  Interventions: Diagnostic Test: PCL COV05 - COVID 19 Ag Rapid FIA test (Rapid Antigen Test)

INTERVENTIONS:
Diagnostic Test: PCL COV05 - COVID 19 Ag Rapid FIA test (Rapid Antigen Test) — The PCL COV05 - COVID 19 Ag Rapid FIA test has FSC and CE approvals for the qualitative detection of SARS-CoV-2 Antigens from human oropharyngeal swabs and deep sputum samples. The manufacturer is PCL Corporation Ltd 17F, 128 B-dong, Courthouse-ro, Songpa-gu, Seoul, South Korea.

SUMMARY:
This study is to evaluate the utility of the PCL Rapid Antigen Test for Coronavirus (COVID-19) in a real world clinical setting. The PCL test has completed laboratory validation and holds a European CE marking for in vitro diagnostic devices. These tests have been made available to South West Pathology Services as a donation in kind by iPP (Integrated Pathology Partnership). They have been widely used in South Korea.

This study will test the practical delivery of the test in terms of time constraints and error rates. We will also compare the objective performance to the current standard diagnostic test for COVID-19 and against a proven serological antibody test when a suitable reference testing becomes available.

We will recruit patients having a SARS CoV-2 PCR swab test and ask for consent to test them with the PCL antigen test in parallel. We aim to study 200 patients split across three sites; Musgrove Park Hospital, Basildon University Hospital and Southend University Hospital. The results will not be used to guide clinical decision making. Patients having a COVID PCR test will be asked to read the patient information sheet and asked if they would like to participate. The patients will be asked to have a second nasal/throat swab taken shortly after their swab for the PCR test.

Written informed consent will be taken for whole blood or plasma left over from any routine clinical sample to be stored as anonymised samples for future testing once a reference test becomes available.

We will report results of the onsite clinical diagnostic test and the PCL antigen test with the number of the kit used, and test date. Anonymised information about year of birth, gender and place of testing will be collected alongside date of onset, symptoms and immunodeficiency status or significant conditions.

DETAILED DESCRIPTION:
Participants will be identified as they attend assessment areas or testing facilities hosted by the recruiting NHS centres. They will be screened by clinical staff and identified to the research team.

Consent will be taken by a clinical staff member or research staff member with the aim of reducing the number of contacts with the patients and minimising the usage of personal protective equipment.

The consent form gives the patient the opportunity to ask further questions. Only those that are able to consent for themselves will be recruited for this trial.

We want to allow patients as long as possible to make a decision to participate but we feel it is important if possible that the swab samples are taken during the same patient contact (reducing PPE usage and minimising additional staff exposures). However there should not be undue delay to clinical testing therefore we propose if due to clinical urgency potential participants do not have sufficient time to consider the patient information sheet and discuss the trial prior to the PCR swab being taken they can have up to 24 hours to consider this information and participate if they wish to.

Consent will be taken by a clinical staff member or research staff member reducing the number of contacts with the patients. They will then be assigned a trial number used to identify them during the trial. The consent form that will be photocopied and reprinted on clean paper, with the original staying with the patient. The clean copy will be stored in the patient's notes and the case record file.

The current standard COVID PCR swab will be taken and a second swab taken immediately after for use in the rapid antigen test. As the swab process can be uncomfortable after the first swab is taken for the standard clinical test (PCR) the participant's consent will be confirmed again prior to taking the second swab required for the antigen test. After consent the research team will complete an anonymised data case record form from the notes and clinical management database. Participant's year of birth and date of onset of symptoms if symptomatic will be documented.

From routine blood samples taken by phlebotomy or clinical staff consent will be sort to store a leftover sample. This will be processed and stored by research laboratory staff. This will be stored in an anonymised secure research freezer.

In the laboratory their swab for the PCL COVID19 Ag rapid FIA will be run on the test platform. Following the test the swab will be destroyed as per local guidelines for contaminated items. This will performed by dedicated research laboratory scientists. Participant's results from this antigen test will not be used to make clinical decisions. We will not be able to feedback participants' individual results.

Participants are expected to be in the study for total of 20 minutes total although this will be spread over their patient journey so they have sufficient time to read the information leaflet and ask questions.

ELIGIBILITY:
Inclusion Criteria:

* Participant has clinical indication for a COVID diagnostic test and a clinical blood sample from which whole blood or plasma will be leftover for storage

Exclusion Criteria:

* Inability to give written informed consent.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 200 (Estimated)
Dates: Start 2020-06 (Estimated); Primary Completion 2021-06 (Estimated); Study Completion 2021-08 (Estimated)

PRIMARY OUTCOMES:
To compare the result of SARS-COV2 PCR test to PCL rapid antigen test | within 24 hours
  Compare the sensitivity and specificity of the rapid antigen testing to current PCR test and any future developed reference test

SECONDARY OUTCOMES:
Number of technically failed samples due to test issues. | At time of testing (within 30 minutes)
  Number of PCL antigen tests that are invalid (no control testing line)
Time taken for PCL Antigen test result | within 30 minutes
  Time from swab being taken to result being read by point of care analyser, manufacturer anticipates 10-15 minutes

CONTACTS AND LOCATIONS:
Locations (1):
- Musgrove Park Hospital, Taunton, Somerset, United Kingdom

IPD SHARING:
Plan to Share IPD: Yes
anonymised individual data would be available to be shared on request from other research teams/public health bodies but no formal plans in place at time of submission
Supporting Information: Study Protocol, CSR
Time Frame: on study completion and for 5 years after
Access Criteria: other clinical researchers or public health bodies evaluating diagnostic tests for COVID-19